CLINICAL TRIAL: NCT02808975
Title: A Phase 4, Double-blind, Randomized, Placebo-Controlled, Multicenter Study to Assess the Safety and Efficacy of Adalimumab Used in Conjunction With Surgery in Subjects With Moderate to Severe Hidradenitis Suppurativa
Brief Title: Safety and Efficacy of Adalimumab (Humira) for Hidradenitis Suppurativa (HS) Peri-Surgically
Acronym: SHARPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M15-574; 2015-005161-23 (EudraCT Number)
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Results first posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: Hidradenitis Suppurativa; Axilla; Inguinal region; Hurley Stage I, II, or III; Adalimumab; Secondary intention; Abcess and inflammatory nodule (AN) count
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Period A: Day 1- 4 subcutaneous (SC) injections; Week 2- 2 SC injections; Weeks 4-12- 1 SC injection each week
  Period B: Weeks 13-14- 1 SC injection each week
  Period C: Weeks 15-23- 1 SC injection each week
  Interventions: Drug: Placebo
- Adalimumab (Active Comparator): Period A: Day 1- 4 subcutaneous (SC) 40 mg injections; Week 2- 2 SC 40 mg injections; Weeks 4-12- 1 SC 40 mg injection each week
  Period B: Weeks 13-14- 1 SC 40 mg injection each week
  Period C: Weeks 15-23- 1 SC 40 mg injection each week
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Placebo — Subcutaneous injections administered as described in arm description
  Arms: Placebo
Drug: Adalimumab — Subcutaneous injections administered as described in arm description
  Other Names: Humira
  Arms: Adalimumab

SUMMARY:
The objective of this study was to assess the safety and efficacy of adalimumab prior to surgery in participants with moderate to severe Hidradenitis Suppurativa (HS) who were surgical candidates.

DETAILED DESCRIPTION:
This was an interventional, randomized, double-blind (DB), placebo-controlled study. The study duration included a 30-day Screening Period, an initial 12-week DB treatment pre-surgery period (Period A), a 2-week peri-operative period with continuation of weekly DB study drug administration (Period B), and a subsequent 10-week DB treatment post-operative period (Period C). Randomization (in a 1:1 ratio) in Period A was stratified by baseline Hurley Stage (II versus III) and anatomical location of the planned surgical site (i.e., axilla versus inguinal region). The projected size of the surgical excision established by the designated surgeon during the Screening Period (calculated from a tracing of the outer perimeter onto an acetate sheet or equivalent) was recorded. In Period B, the designated surgeon measured and recorded the surface area of the actual surgery, with surgery occurring during Week 13. Surgery and post-operative management (e.g., hospitalization, surgical wound care) was per local practice. No study drug was administered at Week 24, the final study visit. Participants were able to begin commercial product (as prescribed by the participants's physician) after all Week 24 procedures were completed.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have skin lesions that are diagnostic of Hidradenitis Suppurativa (HS) for at least 1 year (365 days) prior to the Baseline visit
* Participant must have at least 3 distinct anatomical regions involved with inflammatory (also termed 'active') HS lesions; plus

  * either one axilla or one inguinal region (limited to the inguino-crural fold and adjacent areas) that requires excisional surgery, and
  * with at least one of the other affected HS regions (e.g., contralateral inguinal region, buttocks, inframammary region) rated as Hurley Stage II or III
* Participant must have a total abscess and inflammatory nodule (AN) count of greater than or equal to 3 at the Baseline visit within the HS non-surgical sites
* The HS surgical site must contain at least one active HS lesion
* The HS surgical site must require excisional surgery and is large enough to require healing by secondary intention as assessed by the designated surgeon

Exclusion Criteria:

* Participant has a draining fistula count of greater than 20 at the Baseline visit
* Participant requires surgery at any anatomical site other than an unilateral axilla or inguinal region site
* Participant requires surgical management prior to Week 13
* Participant requires, based on the designated surgeon's assessment, excisional surgery with primary closure as the method of closure being most beneficial for the participant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2016-07-18 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (55):
- United States (9):
  - Wallace Medical Group, Inc. /ID# 171289, Beverly Hills, California
  - Encino Research Center / T. Jo /ID# 171347, Encino, California
  - University of California Irvine /ID# 170054, Irvine, California
  - Tulane Univ /ID# 168441, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center /ID# 168438, Boston, Massachusetts
  - University of Michigan Hospitals /ID# 200667, Ann Arbor, Michigan
  - Univ NC Chapel Hill /ID# 168446, Chapel Hill, North Carolina
  - Penn State Hershey Medical Ctr /ID# 168447, Hershey, Pennsylvania
  - Rhode Island Hospital /ID# 168439, Providence, Rhode Island
- Belgium (2):
  - CUB Hospital Erasme /ID# 150907, Brussels, Brussels Capital
  - UZ Gent /ID# 150906, Ghent, Oost-Vlaanderen
- Canada (2):
  - NewLab Clinical Research Inc. /ID# 151315, St. John's, Newfoundland and Labrador
  - York Dermatology Clinic and Research Centre /ID# 151314, Richmond Hill, Ontario
- Colombia (2):
  - Fundacion Valle Del Lili /ID# 151565, Cali
  - Hospital Pablo Tobon Uribe /ID# 152693, Medellín
- Czechia (2):
  - Fakultni nemocnice Ostrava /ID# 169174, Ostrava, Praha 5
  - Fakult Nem Kralovske Vinohrady /ID# 169173, Prague
- Denmark (2):
  - Bispebjerg Hospital /ID# 150796, Copenhagen NV, Capital Region
  - Sjaellands Universitets Hospit /ID# 150795, Roskilde, Region Sjælland
- France (2):
  - Polyclinique Courlancy /ID# 157761, Reims
  - Hopital Prive d'Antony /ID# 157347, Antony, Île-de-France Region
- Germany (5):
  - Universitaetsklinikum Erlangen /ID# 167251, Erlangen, Bavaria
  - Charité Universitätsmedizin Campus Mitte /ID# 150875, Berlin
  - Klinikum Ruhr Univ Bochum /ID# 150873, Bochum
  - Klinikum Darmstadt GmbH /ID# 150874, Darmstadt
  - Staedtisches Klinikum Dessau /ID# 150876, Dessau
- Greece (3):
  - University General Hospital Attikon /ID# 150841, Athens, Attica
  - Genl Hospital Andreas Syggros /ID# 150840, Athens
  - Genl Hospital Andreas Syggros /ID# 150842, Athens
- St Vincent's University Hosp /ID# 150043, Dublin, Ireland
- Italy (4):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico /ID# 150069, Milan, Lombardy
  - A.O.U Sant'Anna di Ferrara /ID# 150066, Ferrara
  - Universita degli Studi di /ID# 150068, Modena
  - Policlinico Univ Tor Vergata /ID# 150142, Rome
- Hospital Universitario Dr. Jose Eleuterio Gonzalez /ID# 151027, Monterrey, Nuevo León, Mexico
- Netherlands (3):
  - Radboud Universitair Medisch Centrum /ID# 152157, Nijmegen, Gelderland
  - Universitair Medisch Centrum Groningen /ID# 150662, Groningen
  - Erasmus Medisch Centrum /ID# 150672, Rotterdam
- Haukeland University Hospital /ID# 152662, Bergen, Hordaland, Norway
- Prywatny Osrodek Chirurgii Plastycznej Andrzej Bieniek /ID# 169413, Wroclaw, Lower Silesian Voivodeship, Poland
- Centro Hospitalar de Sao Joao, EPE /ID# 150885, Porto, Portugal
- Romania (2):
  - Spitalul Universitar de Urgenta Elias /ID# 151072, Bucharest, București
  - Spitalul Municipal de Urgenta Timisoara /ID# 151073, Timișoara, Timiș County
- Russia (2):
  - City Clinical Hospital 15 /ID# 151281, Moscow
  - NW State Med Univ NA Mechnikov /ID# 151197, Saint Petersburg
- King Faisal Specialist Hospital and Research Centre /ID# 153769, Riyadh, Najran Region, Saudi Arabia
- Spain (5):
  - Corporac Sanitaria Parc Tauli /ID# 150789, Sabadell, Barcelona
  - Hospital Univ Germans Trias I Pujol /ID# 150787, Badalona
  - Hospital Santa Creu i Sant Pau /ID# 152742, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 150788, Madrid
  - Hospital de Manises /ID# 150790, Manises
- Karolinska Univ Sjukhuset /ID# 150817, Solna, Sweden
- Turkey (Türkiye) (2):
  - Hacettepe University Medical Faculty /ID# 150829, Ankara
  - Uludag University Medical Faculty /ID# 150831, Bursa
- Whipps Cross Univ Hospital /ID# 151699, London, London, City of, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Bechara FG, Podda M, Prens EP, Horvath B, Giamarellos-Bourboulis EJ, Alavi A, Szepietowski JC, Kirby J, Geng Z, Jean C, Jemec GBE, Zouboulis CC. Efficacy and Safety of Adalimumab in Conjunction With Surgery in Moderate to Severe Hidradenitis Suppurativa: The SHARPS Randomized Clinical Trial. JAMA Surg. 2021 Nov 1;156(11):1001-1009. doi: 10.1001/jamasurg.2021.3655. PMID 34406349
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Intent-to-Treat (ITT) population: all participants who were randomized at the Baseline visit
Period: Overall Study
Arm/Group | Placebo | Adalimumab
Started | 103 | 103
Completed | 81 | 84
Not Completed | 22 | 19
Not completed — Adverse Event | 3 | 4
Not completed — Withdrew consent | 9 | 8
Not completed — Lost to Follow-up | 4 | 6
Not completed — Planned HS surgery performed prior Wk 13 | 1 | 0
Not completed — Other, not specified | 5 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population: all participants who were randomized at the Baseline visit
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Adalimumab | Total
Number analyzed (Participants) | 103 | 103 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (10.81) | 38.5 (11.71) | 37.6 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 51 | 106
  Male | 48 | 52 | 100
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 97 | 96 | 193
  Black or African American | 4 | 4 | 8
  Asian | 1 | 1 | 2
  American Indian or Alaska Native | 0 | 2 | 2
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  Multiple | 0 | 0 | 0
  Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Hidradenitis Suppurativa Clinical Response (HiSCR) at Week 12
Description: HiSCR is defined as at least a 50% reduction in the abscess and inflammatory nodule (AN) count with no increase in abscess count and no increase in draining fistula count relative to Baseline.
Time Frame: At Week 12
Population: Intent-to-Treat (ITT) population: all participants who were randomized at the Baseline visit; non-responder imputation (NRI) was used for missing data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Adalimumab
Number analyzed (Participants) | 103 | 103
percentage of participants | 34.0 [24.8 to 43.1] | 47.6 [37.9 to 57.2]
Statistical Analysis 1: Comparison: Placebo vs Adalimumab; Test type: Superiority; p = 0.049, Cochran-Mantel-Haenszel; Across all strata, P-value calculated from Cochran-Mantel-Haenszel test adjusted for strata. Stratum containing zero count: 0.1 added to each cell

2. Secondary Outcome: Percentage of Participants Achieving HiSCR-es at Week 12
Description: Hidradenitis Suppurativa Clinical Response-es (HiSCR-es) is defined as at least a 50% reduction in the abscess and inflammatory nodule (AN) count with no increase in abscess count and no increase in draining fistula count relative to Baseline, excluding the Hidradenitis Suppurativa surgical site.
Time Frame: At Week12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Adalimumab
Number analyzed (Participants) | 103 | 103
percentage of participants | 35.0 [25.7 to 44.2] | 47.6 [37.9 to 57.2]
Statistical Analysis 1: Comparison: Placebo vs Adalimumab; Test type: Superiority; p = 0.067, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants Achieving HiSCR-es at Week 24
Description: as for outcome 2
Time Frame: At Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Adalimumab
Number analyzed (Participants) | 103 | 103
percentage of participants | 31.1 [22.1 to 40.0] | 51.5 [41.8 to 61.1]
Statistical Analysis 1: Comparison: Placebo vs Adalimumab; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Percent Change in the Surface Area of the Hidradenitis Suppurativa (HS) Surgical Site From Baseline to Week 12
Description: The projected size of the surgical excision established by the designated surgeon during the Screening Period (calculated from a tracing of the outer perimeter onto an acetate sheet or equivalent) was recorded by the study physician. The change in the surface area of the projected HS surgical site from Baseline to Week 12 was documented.
Time Frame: From Baseline to Week 12
Population: Observed case (OC) analysis was performed on the intent-to-treat (ITT) population. The ITT population consisted of all participants who were randomized at the Baseline visit.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from Baseline
Arm/Group | Placebo | Adalimumab
Number analyzed (Participants) | 79 | 76
percent change from Baseline | 26.233 [-31.684 to 84.150] | 68.190 [8.485 to 127.896]
Statistical Analysis 1: Comparison: Placebo vs Adalimumab; Test type: Superiority; p = 0.313, ANCOVA; Across all strata, P-values are calculated from ANCOVA with stratum, baseline value, and treatment in the model

5. Secondary Outcome: Percentage of Participants at Week 12 That Require a Less Extensive Surgery Than the Surgical Plan (Determined at Baseline) or No Surgery
Description: The projected size of the surgical excision established by the designated surgeon during the Screening Period (calculated from a tracing of the outer perimeter onto an acetate sheet or equivalent) was recorded by the study physician. The change in the surface area of the projected HS surgical site from Baseline to Week 12 was documented, and the percentage of participants at Week 12 requiring a less extensive surgery than the surgical plan (determined at Baseline) or no surgery as determined by the designated surgeon was recorded.
Time Frame: At Week 12
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Adalimumab
Number analyzed (Participants) | 87 | 82
percentage of participants | 43.7 [33.3 to 54.1] | 46.3 [35.5 to 57.1]
Statistical Analysis 1: Comparison: Placebo vs Adalimumab; Test type: Superiority; p = 0.746, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the first dose of study drug until 70 days after the last dose of study drug, up to 33 weeks.
Description: TEAEs and SAEs are defined as any adverse event (AE) with an onset date that is on or after the first dose of study drug until 70 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Placebo | Adalimumab
All-Cause Mortality (participants affected / at risk) | 0/103 | 2/103
Serious Adverse Events (participants affected / at risk) | 3/103 | 7/103
Other Adverse Events (participants affected / at risk) | 43/103 | 48/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=103) | Adalimumab (N=103)
CARDIOVASCULAR DISORDER (Cardiac disorders) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
BLASTOCYSTIS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
TESTIS CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
RUPTURED CEREBRAL ANEURYSM (Nervous system disorders) | 0 (0) | 1 (1)
HIDRADENITIS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=103) | Adalimumab (N=103)
DIARRHOEA (Gastrointestinal disorders) | 4 (4) | 6 (6)
NASOPHARYNGITIS (Infections and infestations) | 19 (24) | 19 (23)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 8 (9) | 14 (14)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)
DIZZINESS (Nervous system disorders) | 6 (7) | 2 (2)
HEADACHE (Nervous system disorders) | 14 (29) | 13 (13)
HIDRADENITIS (Skin and subcutaneous tissue disorders) | 15 (19) | 14 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/75/NCT02808975/SAP_000.pdf
  • Study Protocol (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT02808975/Prot_001.pdf